CLINICAL TRIAL: NCT05576688
Title: Investigation of the Relationship Between Trunk Control and Balance, Gait, Functional Mobility and Fear of Falling in People With Alzheimer's Disease
Brief Title: Trunk Control, Balance, Gait, Functional Mobility and Fear of Falling in People With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 2022/30/09
Record Dates: First submitted 2022-09-30; First posted 2022-10-12 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Physical Therapy
Keywords: trunk control; balance; gait; functional mobility; fear of falling
MeSH Terms: interventions — Gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alzheimer's disease (Experimental): People with Alzheimer's disease who were diagnosed with Alzheimer's disease according to NINCDS/ARDRA diagnostic criteria by a neurologist and whose cognitive level was between 18-23 points according to Mini Mental State Examination.
  Interventions: Other: Balance; Other: Trunk control; Other: Gait; Other: Functional mobility; Other: Fear of falling
- Healthy older adults (No Intervention): 33 healthy older adults with matching ages and gender.

INTERVENTIONS:
Other: Balance — Balance was evaluated with Berg Balance Scale (BBS), Functional Reach Test (FRT), One Leg Stance Test (OLST) and Five-Repeat Sit-and-Stand Test (5STS). BBS consists of 14 functional tasks of increasing difficulty, each scored on a scale ranging from 0 to 4. The maximum possible score is 56, indicating no identifiable balance difficulties. FRT measures the maximum distance that participants can reach forward with their dominant arm raised to 90 degrees without moving their feet, which were positioned 10 cm apart. OLST measures the time one is able to stand on one lower limb without support. The test was repeated for both sides. 5STS assesses the time it takes to get up and sit from the chair five times. Measurements were repeated 3 times and the average duration was calculated as a patient score.
  Arms: Alzheimer's disease
Other: Trunk control — Trunk control was evaluated with Trunk Impairment Scale (TIS).TIS evaluates static sitting balance, dynamic sitting balance, and trunk coordination on a scale from 0 to 23 points, a higher score indicating a better performance.
  Arms: Alzheimer's disease
Other: Gait — Gait was evaluated with Dynamic Gait Index (DGI). DGI has 8 items: walking, walking while changing speed, walking while turning the head horizontally and vertically, walking with pivot turn, walking over and around obstacles, and stair climbing. The scoring of the DGI is based on a 4-point scale ranging from 0 to 3, with 0 indicating severe impairment and 3 indicating normal ability. The best performance total score is 24. A low composite DGI score indicates greater impairment in gait.
  Arms: Alzheimer's disease
Other: Functional mobility — Functional mobility was evaluated with Timed Up and Go Test (TUG). TUG is a test of the time required for an individual to stand up from a chair with armrests, walk 3 m, turn, walk back to the chair, and sit down. The stopwatch timing started when the participant's bottom left the chair and ended when the bottom made contact with the chair after the walk.
  Arms: Alzheimer's disease
Other: Fear of falling — Fear of falling was evaluated with the Falls Efficacy Scale-International (FES-I). FES-I was used to assess the level of concern about falls during 16 activities of daily living, ranging from basic to more demanding activities including social activities that may contribute to quality of life. It was administered as a self-report questionnaire.
  Arms: Alzheimer's disease

SUMMARY:
The purposes of this study were to investigate the relationship between trunk control and balance, gait, functional mobility, and fear of falling in people with Alzheimer's disease and to compare trunk control, balance, gait, functional mobility, and fear of falling in people with Alzheimer's disease and healthy older adults.

Balance, an essential motor skill necessary to perform both static and dynamic everyday activities with stability and security, is impaired in people with Alzheimer's disease when compared to cognitively preserved elderlies. Gait and functional mobility disorders are also observed in people with Alzheimer's disease from the early period of the disease. People with Alzheimer's disease tend to fall more often and are more seriously injured from falls than cognitively intact older adults. The annual incidence rate for falling is 60% to 80% for older adults with Alzheimer's disease, over twice the incidence of age-matched cognitively intact older adults.

Trunk control is shown among the most important factors that ensure the balance and walking of the individual in different environments and conditions during functional activities. Optimal trunk control relies on adequate somatosensory, motor, and musculoskeletal systems, which are frequently compromised in people with Alzheimer's disease. For this reason, the investigators think that trunk control may be affected in people with Alzheimer's disease compared to healthy older adults and may be related to balance, gait, functional mobility and fear of falling.

DETAILED DESCRIPTION:
The study was carried out with the purpose of investigating the relationship between trunk control and balance, gait, functional mobility, and fear of falling in people with Alzheimer's disease and comparing trunk control, balance, gait, functional mobility, and fear of falling in people with Alzheimer's disease and healthy older adults.

35 people with Alzheimer's disease and 33 healthy older adults with matching ages and genders were included the study. Trunk control with Trunk Impairment Scale; balance with Berg Balance Scale, Functional Reach Test, One-Leg Standing Test and Five-Repeat Sit-and-Stand Test; gait with Dynamic Gait Index; functional mobility with Timed Up and Go Test; fear of falling with Falls Efficacy Scale-International were evaluated.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of Alzheimer's disease according to the NINCDS/ARDRA diagnostic criteria by a neurologist.
* Having a cognitive level between 18-23 points according to the Mini Mental Status Examination.
* Must be able to walk independently with and/or without assistive device.

Exclusion Criteria

* Having a history of cerebrovascular disease, epilepsy and brain tumor.
* Having a cognitive level below 18 points according to the Mini Mental Status Examination.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Trunk control | 1 month
  Trunk control was evaluated with Trunk Impairment Scale (TIS). TIS evaluates static sitting balance, dynamic sitting balance, and trunk coordination on a scale from 0 to 23 points, a higher score indicating a better performance.

SECONDARY OUTCOMES:
Functional balance | 1 month
  Functional balance was evaluated with Berg Balance Scale (BBS). BBS consists of 14 functional tasks of increasing difficulty, each scored on a scale ranging from 0 to 4 (0: unable to perform the task; 4: task is performed independently). The maximum possible score is 56, indicating no identifiable balance difficulties.
Dynamic bilateral stance balance | 1 month
  Dynamic bilateral stance balance was evaluated with Functional Reach Test (FRT). FRT, a test of dynamic bilateral stance balance. This test measures the maximum distance that participants can reach forward with their dominant arm raised to 90 degrees without moving their feet, which were positioned 10 cm apart. The distance of additional reach from the starting position was recorded (in centimeters).
One leg standing balance | 1 month
  One leg standing balance was evaluated with One Leg Stance Test (OLST). OLST measures the time one is able to stand on one lower limb without support. This test is a clinical tool to assess postural steadiness in a static position by quantitative measurement. The participant was asked to stand on one leg for 30 seconds while the knee was in 90° flexion. Two measurements were made with a stopwatch and the best measurement score was recorded. The test was repeated for both sides.
Balance | 1 month
  Balance was evaluated with Five-Repeat Sit-and-Stand Test (5STS). 5STS required a straight-back armless chair of standard height (45cm) placed firmly against a wall. After performing an initial single chair stand with arms folded across the chest and feet flat on the floor, the time to complete 5 repeat chair stands was recorded in seconds. A stopwatch was provided to participants who used a suitable chair in their home for all home-based tests Measurements were repeated 3 times and the average duration was calculated as a patient score.
Gait | 1 month
  Gait was evaluated with Dynamic Gait Index (DGI). DGI has 8 items: walking, walking while changing speed, walking while turning the head horizontally and vertically, walking with pivot turn, walking over and around obstacles, and stair climbing. The scoring of the DGI is based on a 4-point scale ranging from 0 to 3, with 0 indicating severe impairment and 3 indicating normal ability. The best performance total score is 24. A low composite DGI score indicates greater impairment in gait
Functional mobility | 1 month
  Functional mobility was evaluated with Timed Up and Go Test (TUG). TUG is a test of the time required for an individual to stand up from a chair with armrests, walk 3 m, turn, walk back to the chair, and sit down. The stopwatch timing started when the participant's bottom left the chair and ended when the bottom made contact with the chair after the walk.
Fear of falling | 1 month
  Fear of falling was evaluated with the Falls Efficacy Scale-International (FES-I). FES-I is used to assess the level of concern about falls during 16 activities of daily living, ranging from basic to more demanding activities including social activities that may contribute to quality of life. It was administered as a self-report questionnaire. The level of concern for each item was scored on a 4-point scale (1: not at all, 2: somewhat, 3: quite a lot, 4: very), with the total score range being 16 to 64.

CONTACTS AND LOCATIONS:
Overall Officials: Taskin Ozkan, Doctorate, Principal Investigator — Giresun University Vocational School of Health Services Therapy and Rehabilitation Department
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)